CLINICAL TRIAL: NCT03594188
Title: Effects of Serum From Hepatocellular Carcinoma Surgery Patients Under Different Anesthetic Methods on Hepatic Cancer Cell Malignancy in Vitro
Brief Title: Effects of Anesthetic Methods on Hepatic Cancer Cell Malignancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEP201807
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia (Experimental): Patients in this group will have RF ablation for treatment of HCC under general anesthesia.
  Interventions: Procedure: anesthetic methods
- local anesthesia (Active Comparator): Patients in this group will have RF ablation for treatment of HCC under local anesthesia.
  Interventions: Procedure: anesthetic methods

INTERVENTIONS:
Procedure: anesthetic methods — Patients will receive standard GA or LA for RF surgery.

SUMMARY:
Numerous studies found that anesthetic methods can influence the recurrence of tumor and the overall survival of patients after primary cancer surgery. Radiofrequency (RF) ablation is now widely used in clinic for treatment of hepatocellular carcinoma (HCC). Currently, diverse anesthetic methods, including general anesthesia (GA), epidural anesthesia and local anesthesia (LA), are used for RF ablation surgery. Using serum from HCC surgery patients randomized to receive either GA or LA during surgery, we investigated the effects of anesthetic methods on proliferation, migration and metastasis in HepG2 hepatic cancer cells in vitro.

ELIGIBILITY:
Inclusion Criteria:

* patients with a single primary liver tumor of 3cm or smaller, who are scheduled for RF ablation surgery

Exclusion Criteria:

* less than 18 or more than 65 years old;
* ASA Physical Status 4 or greater;
* previous surgery in liver (including radiofrequency ablation);
* severe systemic disease (heart, lung, kidney, or immune system);
* INR>1.5 or platelet count <45,000 cells/mm3;
* a history of addiction to opioids;
* with known extension beyond the liver;
* Child-Pugh Class C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
cell proliferation | 1 hour post-surgery
  HepG2 cells will be cultured with serum from patients undergoing RF ablation under GA or LA for 24h and cell proliferation will be measured

SECONDARY OUTCOMES:
cell migration | 1 hour post-surgery
  HepG2 cells will be cultured with serum from patients undergoing RF ablation under GA or LA and cell migration will be measured
cell metastasis | 1 hour post-surgery
  HepG2 cells will be cultured with serum from patients undergoing RF ablation under GA or LA and cell metastasis will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital affliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided